CLINICAL TRIAL: NCT05357131
Title: Neurophysiological Correlates of Dissociation Induced by Virtual Reality Hypnosis (VRH) and Hypnosis (HYP) in a Healthy Participants.
Brief Title: Neurophysiological Correlates of Dissociation Induced by Virtual Reality Hypnosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Oncomfort (Industry); Biowin (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, Responsible of the Sensation and Perception Research Group, in the GIGA CONSCIOUSNESS department, University of Liege
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: QuDDoS - Phase-I
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: Virtual Reality; Hypnosis; Dissociation
MeSH Terms: conditions — Dissociative Disorders | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Cross-over and within-participant control design.
Masking Description: Methodology of virtual reality hypnosis prevents masking the participants and the experimenter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Volunteers - Hypnosis without VR (HYP ) (Experimental): Cross-over and within-participant control design: Participants will receive recorded hypnosis without VR.
  Interventions: Behavioral: Hypnosis without VR (HYP)
- Healthy Volunteers - Hypnosis with VR (VRH) (Experimental): Cross-over and within-participant control design: Participants will receive hypnosis with VR.
  Interventions: Device: Hypnosis with VR (VRH)

INTERVENTIONS:
Behavioral: Hypnosis without VR (HYP) — HYP will last for 15 minutes including an induction phase of 5 minutes. The hypnotic audio script "Heaven of Peace" developped/recorded by Pr. M-E. Faymonville will be used.
  Arms: Healthy Volunteers - Hypnosis without VR (HYP )
Device: Hypnosis with VR (VRH) — The VRH intervention will use the Aqua video session developed by Oncomfort.
  Arms: Healthy Volunteers - Hypnosis with VR (VRH)

SUMMARY:
Hypnosis and virtual reality are potential tools in treating acute pain. Nevertheless, the neurophysiological correlates of such tools used together, i.e. 'virtual reality hypnosis' (VRH) (Patterson et al., 2004) remain mostly understudied. This study aims to improve our knowledge and understanding of the dissociation (i.e., a mental separation of components of behaviours that normally would be processed together) occurring during VRH. This is a randomized controlled study that will be conducted on healthy participants. As the final goal is to propose such a tool in the clinical context, a clinical application will also be carried out subsequently.

Thus the principal outcome is to study dissociation in the context of VRH from a behavioral and neurophysiological point of view.

Secondary objectives aim at identifying factors that influence the dissociative effect seen in VRH, as well as measuring traits of hypnotisability, absorption, immersive abilities, dissociation trait and state, pain, and anxiety levels that might impact the effectiveness of such a tool.

DETAILED DESCRIPTION:
The protocol will follow the following steps:

1. Before the experiment:

   * A medical screening of the medical history and of any concomitant medications will be performed to eligibility.
   * The 6-item Elkins Hypnotisability Scale (EHS) will be used to assess participant hypnotisability.
   * Questionnaire sur la Propension à l'Immersion (QPI) will be used to assess participant immersion tendency.
2. Experimental session: Cross-over and within-participant control design i. Visual Analogue Scale (VAS) :

   * Anxiety.
   * Pain. ii. EEG Resting-state (5-Min.). iii. EEG VRH or EEG Hypnosis alone (HYP) (15-Min.). iv. Adverse Events (AE) during the protocol will be recorded. v. Narrative recording. vi. VAS :
   * Dissociation
   * Absorption
   * Pain
   * Anxiety
   * Arousal/wakefulness
   * Automaticity vii. Time perception (open question) viii. CyberSickness (CSQ) (only if VRH) ix. Presence Questionnaire x. Satisfaction questionnaire xi. Washout Phase (30-Min.) during which we will administer :
   * Six-item State-Trait Anxiety Inventory (STAI-6) .
   * Tellegen Absorption Scale .
   * Dissociative Experience Scales (DES) . xii. VAS:
   * Anxiety
   * Pain xiv. Adverse Events during the protocol will be recorded. xv. Narrative recording. xvi. EEG HYP or EEG VRH Phase (15-Min.). xvii. VAS:
   * Dissociation
   * Absorption
   * Pain
   * Anxiety
   * Arousal/wakefulness
   * Time perception xviii. CSQ (only if VRH) xix. Presence Questionnaire. xx. Satisfaction Questionnaire .

ELIGIBILITY:
Inclusion Criteria: Subject more than 18 years old and equal or less than 65 years old.

Exclusion Criteria:

1. Low auditory and/or visual acuity precludes the use of the device.
2. Head or face wounds precluding the use of the device.
3. Schizophrenia, dissociative disorder or any other psychiatric disorder.
4. Non-proficiency in French (Research language).
5. Patient under 18 years old.
6. Phobia of deep water.
7. Allergy to cutaneous electrodes.
8. Chronic pain and/or chronic analgesics consumption.
9. Medication affecting the autonomic nervous system.
10. Dizziness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Dissociation state | During the procedure
  Corresponds to a dissociation between the bodily sensations and the actual environment that one feels in a particular situation. will be assessed with a numerical rating scale (0= no dissociation; 10 = dissociation from environment).

SECONDARY OUTCOMES:
Dissociation trait | During the procedure
  The amount of dissociation one experiences in one's daily life. Will be assessed with the Dissociative Experience Scale, the higher the score, the more one experiences dissociation in one's daily life.
Hypnotisability | During the procedure
  The susceptibility one has concerning hypnosis. Will be assessed with the Elkins Hypnotizability Scale.
  A score :
  0-3 : low hypnotizability 4-7: medium hypnotizability 8-11 : high hypnotizability 12 : very high hypnotizability
Absorption trait | During the procedure
  The tendency to become fully involved in a perceptual, imaginative or ideational experience. Will be assessed with the Tellegen Absorption Scale, the higher the score the higher the absorption in the daily life.
Anxiety trait | During the procedure
  Level of anxiety one experiences in one's daily life. Will be assessed with the STAI-6 questionnaire. The higher the score, the higher the anxiety one feels in one's daily life.
Immersion propensity (trait) | During the procedure
  Immersion propensity is the amount of sensory input the virtual reality system creates. Will be assessed with the Immersion Propensity questionnaire. The higher the score, the more one is immersed in the virtual environments.
Anxiety state | During the procedure
  The amount of anxiety one experiences in a particular situation. Will be assessed with a visual analogy scale. a score = 0 means no anxiety at all, while a score = 10 means most anxiety ever felt.
Absorption state | During the procedure
  The amount of absroption one experiences in a particular situation. Will be assessed with a numercial rating scale, 0 = no absorption; 10 = fully absorption by the experience.
Pain intensity | During the procedure
  The amount of pain one experiences in a particular situation. Will be assessed with a visual analogy scale, 0= no pain at all; 10= worst pain imaginable.
Automaticity | During the procedure
  A non-voluntary response related to the content of a communication that is intended to be a suggestion. Will be assessed with a numerical rating scale : 0= perfect control; 10 = passive witness.
Arousal/wakefulness | During the procedure
  The amount of arousal one experiences in a particular situation. Will be assessed with a visual analogy scale, 0=not aroused, awaked; 10 = completely aroused, awake.
Time perception | During the procedure
  Open-ended question about one's impression of the duration of the VHR and HYP sessions.
Cybersickness | During the procedure
  Assesses the sickness one might experience after the VRH. Will be assessed with the Cybersickness questionnaire. The higher the score, the more one has experience sickness during the VRH.
Presence | During the procedure
  Refers to the degree to which the subject experiences being in the virtual environment. Will be assessed with the presence questionnaire, the higher the score the higher one has the feeling of really being in the virtual environment.
Satisfaction of the participant | During the procedure
  Assesses the overall satisfaction one has had with the VRH and HYP session. Will be assessed by a self-made satisfaction questionnaire, the higher the score, the more one is satisfied with the experience.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey VANHAUDENHUYSE, PhD, Principal Investigator — CHU of Liège
Locations (1):
- CHU of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No